CLINICAL TRIAL: NCT00301548
Title: Primary Chemotherapy Combined With Perioperative Chemotherapy In Operable Breast Cancer
Brief Title: Perioperative Chemotherapy After Primary Chemotherapy for Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO S31/499
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2006-03-13 (Estimated); Status verified 2006-01

CONDITIONS: Breast Neoplasms; Carcinoma
Keywords: antineoplastic protocols; neoadjuvant therapy; perioperative chemotherapy; fluorouracil
MeSH Terms: conditions — Breast Neoplasms; Carcinoma

INTERVENTIONS:
Drug: perioperative chemotherapy

SUMMARY:
The role of early timing of adjuvant chemotherapy was postulated to be particularly important for patients with endocrine non-responsive disease. The role of cytotoxicity during the period of breast surgery itself and immediately after (perioperative chemotherapy) remained unknown. We investigated in a randomized trial the role of perioperative chemotherapy in patients treated with a preoperative chemotherapy for locally advanced breast cancer and compare it to the preoperative chemotherapy without additional cytotoxic therapy during and immediately after definitive surgery. Patients with T2-3 N0-2 M0 breast cancer, with both estrogen receptors (ER) and progesterone receptors (PgR) expressed in less than 20% of tumor cells, or with absence of progesterone receptors, received up to 6 courses of primary systemic therapy with epirubicin 25 mg/m2 intravenously (i.v.) on days 1 and 2, cisplatin 60 mg/m2 i.v. on day 1, and 5-fluorouracil 200 mg/m2 i.v. daily as continuous infusion (ECF). Patients achieving a partial or complete remission were randomized to continue the infusion of fluorouracil until 2 weeks after surgery (perioperative treatment arm) or to stop fluorouracil infusion one week before surgery, on day 21 of the sixth cycle (control arm).

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer histologically proven > 2 cm, ER and PgR <20% or Any ER and PgR absent (T2,T3 N0-2, M0)
* No treatment with previous chemotherapy/hormonotherapy
* Performance status 0-2 (ECOG scale, Appendix 2)
* Measurable or evaluable lesions
* Age between 18-70 years
* No significant intercurrent illness such as diabetes, cardiovascular, renal or neurologic impairments
* Absence of psychiatric illness
* WBC > 4,000/mm3; PLTS > 100,000/mm3
* AST, ALT, LDH, gamma-GT < 2.5 x upper limit of normal and bilirubin < 3 mg/100 ml
* Informed consent obtained
* Pregnancy test (in fertile women). An effective contraceptive method must be utilized by fertile women.
* Baseline examinations (chest X ray, CT scan, ECG etc) performed within one month prior initiation to therapy

Exclusion Criteria:

* Uncontrolled infection and metabolite disease
* Distant metastases
* Active peripheric and/or central neurological disease
* Active cardiac disease defined as CHF (NYHA III-IV) significant arrhytmias, bilateral bundle branch block or recent (less than 3 months) history of myocardial infarction
* History of second malignancy (exception in situ carcinoma of the uterine cervix and basal or squamous cell carcinoma of the skin)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172
Dates: Start 2000-02; Study Completion 2005-06

PRIMARY OUTCOMES:
Reduction in Ki-67 labeling index

SECONDARY OUTCOMES:
Pathological complete remission rate
Disease-free survival
Toxicity and safety

CONTACTS AND LOCATIONS:
Overall Officials: Colleoni A Marco, MD, Principal Investigator — European Institute of Oncology

REFERENCES:
- [Background] Clahsen PC, van de Velde CJ, Goldhirsch A, Rossbach J, Sertoli MR, Bijnens L, Sylvester RJ. Overview of randomized perioperative polychemotherapy trials in women with early-stage breast cancer. J Clin Oncol. 1997 Jul;15(7):2526-35. doi: 10.1200/JCO.1997.15.7.2526. PMID 9215821
- [Background] Colleoni M, Gelber S, Coates AS, Castiglione-Gertsch M, Gelber RD, Price K, Rudenstam CM, Lindtner J, Collins J, Thurlimann B, Holmberg SB, Cortes-Funes H, Simoncini E, Murray E, Fey M, Goldhirsch A; International Breast Cancer Study Group. Influence of endocrine-related factors on response to perioperative chemotherapy for patients with node-negative breast cancer. J Clin Oncol. 2001 Nov 1;19(21):4141-9. doi: 10.1200/JCO.2001.19.21.4141. PMID 11689582
- [Background] Ludwig Breast Cancer Study Group. Prolonged disease-free survival after one course of perioperative adjuvant chemotherapy for node-negative breast cancer. N Engl J Med. 1989 Feb 23;320(8):491-6. doi: 10.1056/NEJM198902233200804. PMID 2644533